CLINICAL TRIAL: NCT01947062
Title: Evaluation of the Benefits of Oral Metronomic Cyclophosphamide in Combination With Standard Cisplatin-etoposide Based Chemotherapy for Squamous Cell Lung Carcinoma
Brief Title: Metronomic Cyclophosphamide in Combination With Standard Chemotherapy for Squamous Cell Lung Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Swami Rama Cancer Hospital and Research Institute (Industry)
Responsible Party: Principal Investigator, Swaroop Revannasiddaiah, Assistant Professor, Radiotherapy & Clinical Oncology, Swami Rama Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MetroCyclo1
Record Dates: First submitted 2013-09-10; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Lung Cancer; Squamous Cell Carcinoma of the Lung; Locally Advanced and Metastatic Squamous Cell Carcinoma of the Lung
Keywords: NSCLC; Metronomic chemotherapy; Metronomic cyclophosphamide
MeSH Terms: conditions — Lung Neoplasms | interventions — Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard intravenous chemotherapy (Active Comparator): Patients will receive standard intravenous chemotherapy based on cisplatin and etoposide.
  Interventions: Drug: Intravenous Cisplatin & etoposide
- Intravenous with metronomic chemotherapy (Experimental): Patients will receive both intravenous (cisplatin and etoposide based) and metronomic chemotherapy (with oral cyclophosphamide).
  Interventions: Drug: Intravenous Cisplatin & etoposide along with oral cyclophosphamide

INTERVENTIONS:
Drug: Intravenous Cisplatin & etoposide — Patients will receive standard intravenous cisplatin and etoposide based chemotherapy, for a total of six cycles, delivered at three-weekly intervals. In each cycle, the dose of cisplatin will be at 50mg/m2 on days 1 & 2. The dose of etoposide will be 100mg/m2 on days 1, 2 & 3.
  Other Names: Control arm; Standard intravenous chemotherapy
  Arms: Standard intravenous chemotherapy
Drug: Intravenous Cisplatin & etoposide along with oral cyclophosphamide — Patients will be treated with oral cyclophosphamide at a daily dose of 50mg. Patients will also receive standard intravenous cisplatin and etoposide based chemotherapy, for a total of six cycles, delivered at three-weekly intervals. In each cycle, the dose of cisplatin will be at 50mg/m2 on days 1 & 2. The dose of etoposide will be 100mg/m2 on days 1, 2 & 3.
  Other Names: Experimental arm; Intravenous with metronomic chemotherapy
  Arms: Intravenous with metronomic chemotherapy

SUMMARY:
Treatment of locally advanced and metastatic squamous cell carcinoma of the lung involves the use of chemotherapy as the therapeutic mainstay. Platinum-etoposide regimens (such as cisplatin-etoposide) are the most commonly used chemotherapeutic regimen, which is delivered intravenously in the standard three-weekly intervals.

Recent interest in oral metronomic chemotherapy has arisen, especially due to its beneficial effects in delaying disease progression among heavily pre-treated patients with various malignancies.

This study attempts to combine the use of metronomic chemotherapy concurrently during standard intravenous chemotherapy.

DETAILED DESCRIPTION:
Adenocarinoma and squamous cell carinoma are the two major types of non-small cell lung carcinoma. While patients with adenocarcinoma of the lung have the feasibility of treatment with tyrosine kinase inhibitors, the patients with squamous cell carcinoma can only be treated with standard chemotherapy due to the ineffectiveness of tyrosine kinase inhibitors. Thus, the current standard is to treat patients of squamous cell lung cancers with standard intravenous chemotherapy, which is mostly delivered once in three weeks.

Metronomic chemotherapy, meaning the delivery of low doses of chemotherapy, often by an oral approach, on a daily basis so as to maintain a low but definite level of the chemotherapy has received great interest in recent times due to its beneficial effects in terms of extending progression free survival among patients of various malignancies, even after failure with previous conventional therapies. Metronomic chemotherapy is proposed to be active by alternate mechanisms, such as the predominant anti-angiogenic effect, in contrast to the cytotoxic and genotoxic effects of standard chemotherapy.

Metronomic chemotherapy with oral cyclophosphamide has been shown to extend progression free survival when used as a single agent in various malignancies. Given the fact that progression after varying time spans is a rule (rather than the exception) among patients of squamous cell lung cancer being treated with conventional chemotherapy, we have intended to combine the use of oral metronomic chemotherapy given concurrently with standard intravenous cisplatin-etoposide based chemotherapy. We intend to observe a prolongation of progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven squamous cell carcinoma of the lung
* Surgically unresectable or metastatic disease

Exclusion Criteria:

* Severe life limiting diabetes, hypertension or cardiac co-morbidities
* Co-existing tuberculosis
* Brain metastases at presentation
* Non-consenting patients
* Previously treated with any regimen of chemotherapy for existing or previous malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months on average

SECONDARY OUTCOMES:
Response rate | 12 months on average

CONTACTS AND LOCATIONS:
Locations (1):
- Swami Rama Cancer Hospital & Research Institute, Haldwani, Nainital, Uttarakhand, India